CLINICAL TRIAL: NCT02571491
Title: Assessment of the Analgesic Efficacy and Tolerability of the Perioperative Association of the Ketamine With Opiates After Posterior Vertebral Fusion Surgery in Children With Idiopathic Scoliosis
Brief Title: Comparison of the Efficacy of Ketamine in Pediatric Patients With Idiopathic Scoliosis After Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FSJD-ESCOKETA-2010; 2011-000407-41 (EudraCT Number)
Record Dates: First submitted 2015-09-28; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Progressive Infantile Idiopathic Scoliosis
MeSH Terms: interventions — Ketamine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine Hydrochloride (Experimental): Received a combination of ketamine, remifentanil and morphine hydrochloride established by the following dosage regimen:
  * KETAMINE HYDROCHLORIDE 0,5mg/Kg Intravenous bolus administered during the anesthetic induction, followed by 2 mcg / Kg / min of intravenous infusion during and after surgery until 72 hours postoperation
  * during surgery remifentanil 0,3 mcg / kg / min.
  * at the end of the operation morphine hydrochloride150 mcg / kg, PCA infusion postoperatively.
  Interventions: Drug: Ketamine Hydrochloride; Drug: Remifentanil; Drug: Morphine hydrochloride
- Placebo (Placebo Comparator): Received a combination of physiological serum, remifentanil and morphine hydrochloride established by the following dosage regimen:
  * 0,9 % physiological serum 0,5mg/Kg administered by an intravenous (IV) line during the anesthetic induction, followed by 2 mcg / Kg / min of intravenous infusion during and after surgery until 72 hours postoperation
  * during surgery remifentanil 0.3 mcg / kg / min.
  * at the end of the operation morphine hydrochloride150 mcg / kg, PCA infusion postoperatively.
  Interventions: Other: Placebo; Drug: Remifentanil; Drug: Morphine hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — 50 mg/ml, IV (in the vein) during surgery operation, followed by IV ketamine hydrocloride perfusion 2mcg/Kg/min before and until 72 hours after operation Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: KETOLAR 50 mg/ml
  Arms: Ketamine Hydrochloride
Other: Placebo — 50 mg/ml, IV (in the vein) during surgery operation, followed by IV placebo perfusion 2mcg/Kg/min before and until 72 hours after operation
  Other Names: 0,9 % physiological serum
  Arms: Placebo
Drug: Remifentanil — at doses of 0.3 mcg / kg / min during and until the end of the surgical operation
Drug: Morphine hydrochloride — at the dose of 150 mcg / kg, 60 minutes before the extubation procedure and until 72 hours after operation by intravenous infusion

SUMMARY:
Comparison of the Efficacy of ketamine measuring the total consumption of morphine in pediatric patients with idiopathic scoliosis

DETAILED DESCRIPTION:
A randomized unicenter clinical trial, parallel, double-blind study, placebo-controlled group.

Involve the participation of Pediatric patients, aged between 11 and 18 years, of both genders, diagnosed with idiopathic scoliosis and posterior spinal fusion surgery candidates included in the Anesthesia Physical Classification System (ASA) 1 or 2 classes.

Both groups received remifentanil at doses of 0.3 mcg / Kg / min before surgical procedure and a bolus of 150 mcg / Kg of morphine hydrochloride, approximately 60 minutes before extubation, followed by PCA morphine hydrochloride administration.

The patients in the experimental group are treated with a combination of ketamine, remifentanil hydrochloride and morphine while the control group will be treated with a combination of saline, remifentanil and morphine hydrochloride.

Treatment of patients in the study is initiated during the induction of anesthesia and ends at the hospital discharge.

The total duration of patient participation in the study is 6 months. During treatment the patients being admitted are monitored at regular intervals, at week 6, after the 3rd month and at 6 months post-intervention to assess the incidence of chronic pain.

The entire study duration is approximately 24 months. The hypothesis of the study is that the combination of subanesthetic doses of ketamine to opioid drugs during the perioperative period reduces central sensitization processes, resulting in lower consumption of postoperative morphine with fewer adverse effects, postoperative faster recovery and less incidence of chronic pain.

The post-operative analgesia is induced by the use of opioids or other analgesics associated with loco-regional techniques. The technique used in the investigators' center is the patient-controlled analgesia (PCA) with the administration of intravenous opioids.

The association of ketamine to opioid treatment could reduce the consumption of these and can be useful in surgery. No clinical trials have been conducted in children with scoliosis, who underwent posterior lumbar fusion surgical procedure, evaluating the efficacy of post-operative association of ketamine to opioid drugs for both intra and post-operative periods.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders diagnosed with idiopathic scoliosis aged between 8 and 18 years old.
2. Patients of both genders diagnosed with idiopathic scoliosis and candidates for vertebral fusion corrective surgery with instrumentation.
3. Patients with ASA 1 or ASA 2.
4. Patients and/or parents/tutors consent to participate in the clinical trial.

Exclusion Criteria:

1. Patients with chronic preoperative pain.
2. Patients with addiction to narcotics.
3. Patients with a history of allergy, contraindication or intolerance to the drugs used.
4. Patients unable to understand the patient-controlled analgesia system.
5. Patients with mental disorders.
6. Reoperated patients.
7. Patients requiring elective postoperative ventilation.
8. Pregnant patients.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Cumulative Consumption of Epidural Morphine at 72h Postoperatively | in the first 72 hours postoperatively
  For the assessment of the related ketamine analgesic efficacy. Cumulative consumption of epidural morphine administered as loading dose, intraoperatively, of 0,3 mcg/kg/min until the surgery operation and 150mcg/Kg of Morphine hydrochloride 60min before extubation

SECONDARY OUTCOMES:
Change From Baseline in Pain Scores (Visual Analogue Scale) | in the first 72 hours after surgery.
  Pain scores at rest and on cough using a 10cm Visual Analogue Scale(0=no pain, 10=worst possible pain for the analgesic efficacy assessment of the association of Ketamine and opiates
Rates of significant adverse events | every 4 hours from the begin until the end of the surgical operation
  To assess the tolerability of the association of ketamine and opiates
Time to oral tolerability | up to 6 months from the end of the surgical operation
  To assess the efficacy of the association of ketamine and opiates, measuring the time needed from the surgery for reaching the oral tolerability
Time to First Postoperative Ambulation | up to 6 months from the end of the surgical operation
  To assess the efficacy of the association of ketamine and opiates, measuring the time needed to being able to walk without assistance within the room or outside the room
Time to postoperative recovery | up to 6 months from the end of the surgical operation
  Post operation period needed for each patient from the end of the surgery until hospital discharge by counting each patient postoperative hospital night admissions
Change From Baseline in Pain by sensorial test using the Voy Frey filament | in the first 72 hours post surgery
  measure of the area of hyperalgesia of the inflamed skin and the length of the incision after 72 post surgery. The filaments is used to provide a range of forces to the skin of a test subject, in order to find the force at which the subject reacts because the sensation is painful.
Change From Baseline in Pain Scores (Visual Analogue Scale) | at week 6 and after 3 and 6 months post surgery.
  Assessment of pain at week 6 and chronic pain after 3 and 6 months post-surgery using the Visual Analogue Scale pain scale
Change From Baseline in neuropathic pain using Douleur Neuropathique en 4 Questions (DN4) questionnaire | at week 6 and after 3 and 6 months post surgery.
  The (DN4) questionnaire is a screening tool for neuropathic pain consisting of interview questions (DN4-interview) and physical tests. Two questions (I and II) were based on the interview of the patient and two questions (III and IV) were based on a standardized clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Marina Perelló Riera, MD, Principal Investigator — Hospital Sant Joan de Déu Servicio de Anestesiología, Reanimación y Tratamiento del Dolor
Locations (1):
- Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Mao J. Opioid-induced abnormal pain sensitivity: implications in clinical opioid therapy. Pain. 2002 Dec;100(3):213-217. doi: 10.1016/S0304-3959(02)00422-0. No abstract available. PMID 12467992
- [Background] Woolf CJ, Salter MW. Neuronal plasticity: increasing the gain in pain. Science. 2000 Jun 9;288(5472):1765-9. doi: 10.1126/science.288.5472.1765. PMID 10846153
- [Background] Angst MS, Koppert W, Pahl I, Clark DJ, Schmelz M. Short-term infusion of the mu-opioid agonist remifentanil in humans causes hyperalgesia during withdrawal. Pain. 2003 Nov;106(1-2):49-57. doi: 10.1016/s0304-3959(03)00276-8. PMID 14581110
- [Background] Schmid RL, Sandler AN, Katz J. Use and efficacy of low-dose ketamine in the management of acute postoperative pain: a review of current techniques and outcomes. Pain. 1999 Aug;82(2):111-125. doi: 10.1016/S0304-3959(99)00044-5. PMID 10467917